CLINICAL TRIAL: NCT00653445
Title: A 6wk Open-Label, Randomised, Multicentre, Phase IIIb, Parallel Group Study to Compare the Safety & Efficacy of Rosuvastatin 40mg in Comb.With Ezetimibe 10mg in Subjects With Hypercholesterolaemia & CHD or Atherosclerosis or a CHD Risk Equiv. (10 yr Risk Score >20%).
Brief Title: Compare the Safety & Efficacy of Rosuvastatin 40mg in Combination With Ezetimibe 10mg
Acronym: EXPLORER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Elisabeth Björk, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3569C00006
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Hypercholesterolemia; Coronary Heart Disease; Atherosclerosis
Keywords: Low density lipoproteins; Hypercholesterolemia; Coronary Heart Disease; Rosuvastatin; Crestor; Ezetimibe
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease; Atherosclerosis | interventions — Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Rosuvastatin 40mg/Ezetimibe 10mg combination therapy
  Interventions: Drug: Rosuvastatin; Drug: Ezetimibe
- 2 (Experimental): Rosuvastatin 40 mg
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — 40mg
  Other Names: Crestor
Drug: Ezetimibe — 10mg
  Other Names: Zetia
  Arms: 1

SUMMARY:
The purpose of this study is to compare 6 weeks of treatment with rosuvastatin alone compared with 6 weeks of treatment of rosuvastatin combined with ezetimibe in achieving low density lipoprotein level goals.

ELIGIBILITY:
Inclusion Criteria:

* A history of CHD or clinical evidence of atherosclerosis or multiple risk factors that confer a high risk as defined in the protocol.
* Fasting LDL-C concentrations at Visit 1 as defined in the protocol.
* Discontinuation of all lipid lowering therapy at Visit 1.

Exclusion Criteria:

* History of statin induced serious side effects, or serious hypersensitivity reaction to other statins.
* Subjects considered to be unstable by the investigator after the following events: a myocardial infarction (heart attack), unstable angina, myocardial revascularisation or another revascularisation procedure or a transient ischaemic attack (TIA) or stroke.
* Severe congestive cardiac failure (as defined by the protocol - Appendix I).
* Subjects awaiting a planned myocardial revascularisation prior to starting the study (i.e. planned prior to visit 1)..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-06; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of rosuvastatin alone with rosuvastatin combined with ezetimibe by measuring fasting low-density lipoprotein cholesterol (LDL-C) levels at baseline and Week 6

SECONDARY OUTCOMES:
To compare the efficacy of rosuvastatin alone with rosuvastatin combined with ezetimibe by measuring fasting blood lipid levels levels at baseline and Week 6
Safety: by measuring adverse events & abnormal laboratory markers to compare safety & tolerability of rosuvastatin alone with rosuvastatin combined with ezetimibe

CONTACTS AND LOCATIONS:
Overall Officials: Christine Ballantyne, MD, Principal Investigator — Centre for prevention of cardiovascular disease, Texas, USA